CLINICAL TRIAL: NCT00001345
Title: Family Studies in Metabolic Diseases and Mineral Metabolism
Brief Title: Studies of Inherited Diseases of Metabolism
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 930127; 93-DK-0127
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Multiple Endocrine Neoplasia
Keywords: Hypercalcemia; Multiple Endocrine Neoplasia (MEN); Familial Hypocalciuric Hypercalcemia; Hyperparathyroidism; Linkage Analysis; Natural History
MeSH Terms: conditions — Multiple Endocrine Neoplasia; Hypercalcemia; Hypocalciuric hypercalcemia, familial, type 1; Hyperparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Members of families that have had relatives diagnosed with a disease of mineral metabolism. Participants will be asked to give blood samples for DNA extraction.

SUMMARY:
Diseases of mineral metabolism such as familial multiple endocrine neoplasia type 1 (FMEN1), familial hypocaliuric hypercalcemia (FHH), familial hyperparathyroidism (FH), and pseudohypoparathyroidism (PHP) are known as hereditary abnormalities. Meaning these conditions are passed from parents to their children through genes. These specific conditions result in abnormal levels of calcium in the blood.

This study was designed to help researchers understand more about the genes that are responsible for these disorders. By learning more about the genetic process involved in hereditary abnormalities, new tests and treatments can be developed.

Subjects for this study will be members of families that have had relatives diagnosed with a disease of mineral metabolism. Participants will be asked to give blood samples for DNA extraction. DNA is the part of cells that carries genetic information.

The DNA will be analyzed and the results given to the subjects. Genetic counseling will be provided to subjects to aid in interpreting their results....

DETAILED DESCRIPTION:
Familial multiple endocrine neoplasia type 1 (MEN1), familial hypocalciuric (or familial benign) hypercalcemia (FHH), hyperparathyroidism - jaw tumor syndrome (HPT-JT), other causes of familial isolated hyperparathyroidism (FIHP), and pseudohypoparathyroidism (PHP) are disorders of metabolism that are generally inherited in an autosomal dominant fashion. MEN1 is characterized by overgrowth and hyperfunction of the parathyroids, anterior pituitary and gastrointestinal endocrine tissue. MEN1, p15, p18, p21, and p27 are identified genes for MEN1- like states. FHH is characterized by a usually benign syndrome sometimes mistaken for typical primary hyperparathyroidism, which may result in unnecessary and unsuccessful parathyroid surgery. The CASR gene for the calcium-sensing receptor of the parathyroid cell is mutated in most FHH kindreds; a minority of kindreds with FHH have mutation of the GNA11 or AP2S1 gene. HPT-JT is a distinctive subtype of familial isolated hyperparathyroidism that has combinations of parathyroid adenoma, parathyroid cancer, jaw tumor, uterus tumor, kidney tumor and kidney cysts. It is caused by mutation of the CDC73/HRPT2 gene. PHP is characterized by parathyroid hormone resistance, and one form is associated with mutations in the gene encoding the alpha subunit of the stimulatory G protein. We are continuing to collect blood and tissue samples from affected and unaffected members of kindreds with known or suspected MEN1, FHH, HPT-JT, FIHP, PHP, and related disorders for the purpose of geneticanalysis and gene identification. In most cases, the procurement of specimens under this protocol will be at an off-site location. Samples will be processed for extraction of DNA and RNA.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

  1. Patient has possible form of familial hyperparathyroidism. Or case is a clinically unaffected first degree relative of such a patient.
  2. The lower age limit to enter a clinically affected minor into the study is >= 4 years old. However, asymptomatic and possibly unaffected cases will not be enrolled, and blood will not be drawn, before age 5 years in MEN1, MEN1-like, HPT-JT, or FIHP kindreds or before age 10 in FHH kindreds.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects for this study will be members of families that have had relatives diagnosed with a disease of mineral metabolism. Participants will be asked to give blood samples for DNA extraction. DNA is the part of cells that carries genetic information. The DNA will be analyzed and the results given to the subjects. Genetic counseling will be provided to subjects to aid in interpreting their results.
Sampling Method: Non-Probability Sample
Enrollment: 969 (Actual)
Dates: Start 1993-08-19 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Evaluation of metabolic diseases | Yearly
  Studies will be focused around forms of hereditary hypercalcemia, MEN1, FHH, HPT-JT, and FIHP as well as other disorders of mineral metabolism like PHP. In doing so, we will test the hypothesis that MEN1 and MEN1-like states develop as a result of a germ line mutation in MEN1 or a CDKI gene, define the mutations present in the affected members of MEN1 kindreds, and assess the frequency of such mutations in patients with apparently sporadic disease.

CONTACTS AND LOCATIONS:
Overall Officials: Smita Jha, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Spiegel AM, Shenker A, Weinstein LS. Receptor-effector coupling by G proteins: implications for normal and abnormal signal transduction. Endocr Rev. 1992 Aug;13(3):536-65. doi: 10.1210/edrv-13-3-536. No abstract available. PMID 1425488
- [Background] Marx SJ, Attie MF, Levine MA, Spiegel AM, Downs RW Jr, Lasker RD. The hypocalciuric or benign variant of familial hypercalcemia: clinical and biochemical features in fifteen kindreds. Medicine (Baltimore). 1981 Nov;60(6):397-412. doi: 10.1097/00005792-198111000-00002. No abstract available. PMID 7311809
- [Background] Chandrasekharappa SC, Guru SC, Manickam P, Olufemi SE, Collins FS, Emmert-Buck MR, Debelenko LV, Zhuang Z, Lubensky IA, Liotta LA, Crabtree JS, Wang Y, Roe BA, Weisemann J, Boguski MS, Agarwal SK, Kester MB, Kim YS, Heppner C, Dong Q, Spiegel AM, Burns AL, Marx SJ. Positional cloning of the gene for multiple endocrine neoplasia-type 1. Science. 1997 Apr 18;276(5311):404-7. doi: 10.1126/science.276.5311.404. PMID 9103196
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1993-DK-0127.html